CLINICAL TRIAL: NCT03989492
Title: Role of the Sympathetic Nervous System in Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristen Metzler-Wilson (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Kristen Metzler-Wilson, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 95771; 1R15AR069912-01A1 (NIH)
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Rosacea
Keywords: autonomic nervous system; skin blood flow; skin sympathetic nerve activity
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autonomic responses to stressors (Experimental): Protocol 1: mental math and handgrip exercise. Protocol 2: systemic stressors and end-organ receptor stimulation. Protocol 3: local heating.
  Interventions: Other: systemic and local stressors

INTERVENTIONS:
Other: systemic and local stressors — Protocol 1: skin sympathetic nerve activity will be measured during mental math and handgrip exercise. Protocol 2: skin end organ responses will be measured at baseline and in response to systemic stressors and end-organ receptor stimulation. Protocol 3: skin end organ responses will be measured at baseline and during local heating.

SUMMARY:
Rosacea is a common skin disorder which causes facial redness and inflammation in about 16 million Americans, from an unknown cause. Many triggers of rosacea symptoms are stressors that affect the sympathetic ("fight or flight") portion of the nervous system, and a recent pilot study suggests there is sympathetic dysfunction in rosacea. This project will benefit patients, clinicians, and basic scientists by increasing our understanding of sympathetic nervous system involvement in rosacea symptoms in order to develop improved treatments for patients with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy males and non-pregnant/non-lactating females with mild to moderate erythematotelangiectactic rosacea, as well as age-sex matched healthy control subjects.

Exclusion Criteria:

* Neurological, cardiovascular, respiratory, metabolic, muscular, or other dermatological disorders
* Current history of alcohol and/or drug abuse
* Known allergies or hypersensitivities to medications/drugs that are used in the protocol
* Current smoking or regular smoking within the last 2 years
* Body mass index > 35 kg/m2
* Medications or supplements which are known to affect neural, cardiovascular, or muscular responses

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Skin blood flow | Immediate (during the single-day study). This study consists of a one-day protocol, during which this outcome is measured.
  laser Doppler flowmetry
Skin sympathetic nerve activity | Immediate (during the single-day study). This study consists of a one-day protocol, during which this outcome is measured.
  microneurography

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Metzler-Wilson, PT, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No